CLINICAL TRIAL: NCT04605666
Title: CD19-Chimeric Antigen Receptor-T2 Cells for CD19 Positive Relapsed/Refractory B Cell Leukemia/Lymphoma
Brief Title: CD19-CAR-T2 Cells for CD19 Positive B Cell Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2020-098; NFEC-2020-098 (Other: Nanfang Hospital-Ethics Committee)
Record Dates: First submitted 2020-10-25; First posted 2020-10-28 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: B Cell Leukemia; B Cell Lymphoma
Keywords: CAR-T
MeSH Terms: conditions — Leukemia, B-Cell; Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T group (Experimental)
  Interventions: Biological: CD19-CAR-T2 Cells

INTERVENTIONS:
Biological: CD19-CAR-T2 Cells — CD19-CAR-T2 T cells will be infused over 10-15 minutes on Day 0.

SUMMARY:
Chimeric antigen receptor T cells (CAR-T cells) has been recognized a promising treatment option for treating B cell derived malignancy. The purpose of this study is to evaluate the efficacy and safety of third-generation anti-CD19 CAR T-cells (CD19-CAR-T2 Cells) in patients with CD19+ relapsed or refractory (r/r) B-cell acute lymphoblastic leukemia (B-ALL) and B-cell Non Hodgkin Lymphoma (B-NHL).

ELIGIBILITY:
Inclusion Criteria:

* Patient with relapsed and/or refractory CD19+ B-cell leukemia or lymphoma
* Eastern Cooperative Oncology Group (ECOG) performance status <2
* ALT/ AST <3 x normal
* Bilirubin < 2.0 mg/dl
* Creatinine < 2.5 mg/dl and less than 2.5x normal for age
* LVEF< 45%
* Accept white blood cell collection
* Provide informed consent

Exclusion Criteria:

* Previous treatment with investigational gene or cell therapy medicine products
* Active hepatitis B , hepatitis C or HIV infection
* Uncontrolled active infection
* Presence of grade 2-4 acute or extensive chronic GVHD
* Any uncontrolled active medical disorder that would preclude participation as outlined.
* Received non-diagnostic purposes major surgery within the past 4 weeks
* Participated in any other clinical study within the past 4 weeks
* Used murine biological products (except blinatumomab), unless it is proved no anti-mouse antibodies exist.
* Pregnancy or breast-feeding women
* Use of prohibited drugs:
* Steroids: Therapeutic doses of steroids must be stopped > 72 hours prior to CD19-CAR-T2 Cells infusion
* Allogeneic cellular therapy: Any donor lymphocyte infusions (DLI) must be completed > 4 weeks prior to CD19-CAR-T2 Cells infusion
* GVHD therapies: Any drug used for GVHD must be stopped > 4 weeks prior to CD19-CAR-T2 Cells infusion
* Any situation that may increase the risk of the test or interfere with the test results

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
ORR | 3 months
  Overall Response Rate includes Complete Remission (CR) and Complete Remission with Incomplete Blood Count Recovery (CRi), as determined by assessments of peripheral blood, bone marrow, CNS symptoms, physical exam (PE) and CSF. The primary endpoint will be based on the IRC assessment. The local investigator's assessed results will be used for sensitivity analysis.

SECONDARY OUTCOMES:
ORR | 6 months
ORR | 12 months
Adverse Events | 12 months
OS | 1 year
  overall survival
DFS | 1 year
  disease-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Qi-fa Liu, MD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] He B, Lin R, Xu N, Qin L, Wang Z, Wang Q, Li X, Wei X, Wei Y, Tang Z, Fan Z, Huang F, Liu X, Sun J, Xuan L, Li P, Zhou H, Liu Q. Efficacy and safety of third-generation CD19-CAR T cells incorporating CD28 and TLR2 intracellular domains for B-cell malignancies with central nervous system involvement: results of a pivotal trial. J Transl Med. 2025 May 27;23(1):594. doi: 10.1186/s12967-025-06608-x. PMID 40426201